CLINICAL TRIAL: NCT05720078
Title: UNIty-Based MR-Linac Guided Adaptive RadioThErapy for High GraDe Glioma-3 (UNITED-3): Applying a Two Phase, Personalized Margin, Reduced Clinical Target Volume Approach
Brief Title: UNIty-Based MR-Linac Guided Adaptive RadioThErapy for High GraDe Glioma-3 (UNITED-3)
Acronym: UNITED-3
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Principal Investigator, Jay Detsky, Assistant Professor of Radiation Oncology, Sunnybrook Health Sciences Centre
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UNITED-3
Record Dates: First submitted 2023-01-06; First posted 2023-02-09 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2024-11

CONDITIONS: Glioblastoma Multiforme, Adult
MeSH Terms: conditions — Glioblastoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Adaptive, two-phase RT (Experimental)
  Interventions: Radiation: Adaptive, two-phase RT

INTERVENTIONS:
Radiation: Adaptive, two-phase RT — Participants in this arm will be treated with an adaptive, two-phase radiation therapy approach

SUMMARY:
The goal of this study is to test whether an adaptive radiation therapy (RT), two-phase approach in participants with glioblastoma impacts local control compared to standard non-adaptive RT approach. The main questions of the study are to see how this adaptive, two-phase RT approach compares to standard RT in terms of:

* Local control
* Overall and progression-free survival
* Patterns of failure
* Toxicity, Neurological Function, and Quality of Life

DETAILED DESCRIPTION:
Glioblastoma (GBM) is a high grade glioma (brain tumor) that is treated with surgery or biopsy followed by radiotherapy (RT) given daily over 6 weeks with or without an oral chemotherapy. Radiation is targeted to the visible residual tumor on magnetic resonance imaging (MRI) images plus a large margin of 15 to 30 mm to account for possible cancer cells outside the visible tumor and for potential growth or shifts in tumor position throughout the prolonged RT course. Standard RT uses MRI to create a reference plan (with large margins) and treats that same volume every day. This exposes a large amount of healthy brain tissue to radiation leading to toxicity and reduced quality of life.

A new technology, the MR-Linac, combines an MRI scanner and a Linac (radiation delivery machine) into one unit. This allows for "adaptive" RT by obtaining an updated MRI scan each day just prior to treatment, adapting the RT plan to take into account any changes in the tumor or the patient's anatomy on that given day. This allows for a smaller (5 mm) margin on the visible tumor as its position can be tracked daily. The goal of this study is to use adaptive RT with small margins with a two-phase approach to test the impact on local control of the visible tumor compared to the large volumes used with standard non-adaptive RT, as well as impacts on neurocognitive function and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Histopathologically confirmed, based on biopsy or surgical resection, glioblastoma, or grade 4 astrocytoma, as defined by the World Health Organization (WHO)
* Deemed clinically appropriate for long course radiation therapy concurrent with systemic therapy
* Biopsy or surgical resection performed ≤ 12 weeks prior to study entry
* Adequate hematological, renal and hepatic functions as defined by the following required laboratory values obtained within 14 days prior to study entry:

  * Absolute granulocyte count (AGC) > 1.5 x 109/L (1,500 cells/mm3)
  * Platelet count > 100x109/L (100,000 cells/mm3)
  * Serum creatinine < 1.5 times the upper limit of normal
  * Total serum bilirubin < 1.5 times the upper limit of normal
  * Alanine Aminotransferase (ALT, or formerly serum glutamic-pyruvic transaminase (SGPT)) < 2.5 times the upper limit of normal
  * and/or aspartate aminotransferase (AST, or serum glutamic-oxaloacetic transaminase (SGOT)) < 2.5 times the upper limit of normal
* Expected survival ≥ 12 weeks
* Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1 or 2
* Able (sufficiently fluent in English) and willing to complete quality of life questionnaires; however, inability to complete the questionnaires will not make the patient ineligible for the study
* Sufficient estimated glomerular filtration rate (eGFR) of ≥ 30 mL / min/1.73 m2 to allow administration of gadolinium-based contrast agent; patients with eGFR < 30 mL/min/1.73 m2 not on dialysis may be allowed on the study after discussion of risks and benefits and approval by study neuroradiologist(s)
* Completed written informed consent
* Patient must be accessible for treatment and follow-up

Exclusion Criteria:

* Contraindications to MRI examination as per standard MRI screening policy
* Contraindication to Gadolinium-based contrast media
* Inability to lie flat in a supine position for at least 30 minutes
* Inability to tolerate immobilization in a head thermoplastic mask
* Patients > 140 kg and/or a circumference > 60 cm
* Prior therapeutic cranial irradiation
* Leptomeningeal dissemination of disease
* History of other malignancies with the exception of adequately treated non-melanoma skin cancer, or curatively treated other solid tumours with no evidence of disease for ≥ 2 years
* Patients with any condition (e.g. psychological, geographical, etc.) that does not permit compliance with the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2028-04-30 (Estimated)

PRIMARY OUTCOMES:
Rate of marginal failure (if 20-80% of the recurrent GTV (rGTV) falls within the 95% isodose line) | Through study completion, anticipated 6-12 months

SECONDARY OUTCOMES:
Overall survival | Through study completion, anticipated 6-24 months
Progression-free survival | Through study completion, anticipated ~5 months
Rate of local control, in accordance with RANO-HGG criteria | Through study completion, anticipated ~5 months
Patterns of failure | Through study completion, anticipated 6-24 months
Rate of toxicity | Through study completion, anticipated 6-24 months
  Assessed using the Radiation Therapy Oncology Group (RTOG) acute toxicity scale, which assesses acute toxicity using a scale of 0-5, and late toxicity using a scale of 1-4. In both scales, a higher score means a worse outcome.
Health-related Quality of Life | Through study completion, anticipated 6-24 months
  Assessed using the European Organisation for Research and Treatment of Cancer (EORTC) QLQ-C30 to measure quality of life
Changes in neurologic function | Through study completion, anticipated 6-24 months
  Assessed through the Neurologic Assessment in Neuro-Oncology (NANO) scale
Adaptive Radiation Dosimetry | 6 weeks
Functional Imaging Kinetics as a Correlate of Treatment Response | Through study completion, anticipated 12-24 months

CONTACTS AND LOCATIONS:
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No